CLINICAL TRIAL: NCT01977716
Title: The Role of Peritonitis in the Loss of Residual Renal Function, Technique Failure and Mortality in Peritoneal Dialysis Patients
Brief Title: Peritonitis and Loss of Residual Renal Function, Technique Failure and Mortality in Peritoneal Dialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Other Study IDs: R-2013-785-069
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-10

CONDITIONS: Loss of Residual Renal Function; Technique Failure in Peritoneal Dialysis
Keywords: Peritonitis; loss of residual renal function; technique survival
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Incident peritoneal dialysis patients: Patients with chronic kidney disease incident to peritoneal dialysis treatment

SUMMARY:
The primary objective is to analyze peritonitis rate and peritonitis bacteriology as risk factors for loss of residual renal function, technique failure and mortality in chronic kidney disease patients.

Secondary objectives are: To know the current rate of peritonitis in peritoneal dialysis population and to understand the bacteriological profile of peritonitis.

To know the rate and risk factors other than peritonitis involved in the loss of residual renal function.

To analyze the utility of alternative diagnostic tests, such as reagent strips, for early detection of peritonitis when traditional tests are not available.

To analyze the simultaneous measurement of serum creatinine and cystatin-C as alternative measurements of peritoneal clearance and residual renal function.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria include: adult patients with signed informed consent given; there should not be selection for age, gender, primary cause of renal disease.

-

Exclusion Criteria:Patients will not be included if they were previously in hemodialysis or received renal transplant. Patients will also be excluded if they are on immunosuppressive therapy, have diagnosis of cancer, or are seropositive for HIV or hepatitis.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients starting PD as the first dialysis treatment will be considered. Recruitment will take place over a six-months period in hospitals belonging to the Instituto Mexicano de Seguro Social. Inclusion criteria include: adult patients with signed informed consent given; there should not be selection for age, gender, primary cause of renal disease. Patients will not be included if they were previously in hemodialysis or received renal transplant. Patients will also be excluded if they are on immunosuppressive therapy, have diagnosis of cancer, or are seropositive for HIV or hepatitis.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Loss of residual renal function | 25 months
Technique (peritoneal dialysis) failure | 25 months
  Shift to hemodialysis

OTHER OUTCOMES:
Death | 25 months

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Investigación Médica en Enfermedades Nefrológicas, Instituto Mexicano del Seguro Social, Mexico City, Mexico City, Mexico